CLINICAL TRIAL: NCT05829876
Title: Comparison of Cardiac Resynchronisation Therapy (CRT) Response Using High Frequency (HF) - ECG or Q-LV Guided Optimisation for Left Ventricular, Pacing Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRK7831
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either the treatment (HF-ECG guided LV pacing site optimisation) or control (Q-LV guided LV pacing site optimisation) arm, employing a 1:1 randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HF-ECG guided LV pacing site optimisation (Experimental): Participants will have the left ventricular pacing site programmed based on the results of HF-ECG mapping to locate the area of latest activation and best pattern of paced resynchronisation.
  Interventions: Other: High Frequency ECG Mapping
- Q-LV guided LV pacing site optimisation (Active Comparator): Participants will have the left ventricular pacing site programmed based on the results of Q-LV measurement to locate the area of latest activation. This is the standard of care method for pacing site optimisation.
  Interventions: Other: Q-LV Measurement

INTERVENTIONS:
Other: High Frequency ECG Mapping — A high frequency ECG map will be performed to assess the optimum left ventricular pacing site.
  Arms: HF-ECG guided LV pacing site optimisation
Other: Q-LV Measurement — Measurement of Q wave on 12 lead ECG to LV stimulus to assess optimum left ventricular pacing site.
  Arms: Q-LV guided LV pacing site optimisation

SUMMARY:
The research aims to compare the response of Cardiac Resynchronisation Therapy (CRT) using HF ECG guided or the conventional method of Q-LV measurement guided optimisation for left ventricular, pacing site.

DETAILED DESCRIPTION:
The study aims to demonstrate that left ventricular (LV) pacing site optimisation using high frequency (HF) ECG improves LV reverse remodeling response to Cardiac Resynchronization Therapy (CRT), compared with Q-LV (Q-wave on the surface ECG to LV Electrogram) measurement after 6 months of treatment.

Participants will be implanted with a Cardiac Resynchronisation Therapy device with either pacemaker or defibrillator function.

The study is a single-Centre, randomized, prospective trial. One hundred and eighty participants will be assigned to either the treatment (HF-ECG guided LV pacing site optimisation) or control (Q-LV guided LV pacing site optimisation) arm, employing a 1:1 randomization. The participants will be followed up for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • Eligible for implantation of a CRT-D device according to published relevant ESC and CCS guidelines;

  * In sinus rhythm;
  * NYHA class II, III or IV
  * Have reviewed, signed and dated an informed consent.
  * Age 18

Exclusion Criteria:

* Previous implant with a pacemaker, an ICD or a CRT device. (except upgrade from single chamber ICD with a fully functional defibrillation lead) not under recall or surveillance);
* Persistent atrial arrhythmias (or cardioversion for atrial fibrillation) within the past month;
* Ventricular tachyarrhythmia of transient or reversible causes such as acute myocardial infarction (MI), digitalis intoxication, drowning, electrocution, electrolyte imbalance, hypoxia or sepsis, uncorrected at the time of the enrolment;
* Incessant ventricular tachyarrhythmia;
* Unstable angina, or acute MI, Coronary Artery Bypass-Grafting (CABG), or Percutaneous Coronary Intervention (PCI) within the past 4 weeks;
* Correctable valvular disease that is the primary cause of heart failure;
* Indication for valve repair or replacement;
* Recent Cerebro-Vascular Accident (CVA) or Transient Ischemic Attack (TIA) (within the previous 3 months);
* On transplant waiting list;
* Previous heart transplant;
* Already included in another clinical study that could confound the results of this study;
* Life expectancy less than 1 year;
* Inability to understand the purpose of the study;
* Unavailability for scheduled follow-up or refusal to cooperate;
* Age of less than 18 years;
* Pregnancy;
* Drug addiction or abuse;
* Under guardianship.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Reverse Remodelling | 6 months
  Absolute difference in left ventricular end systolic volume greater than or equal to 10%

SECONDARY OUTCOMES:
Change in NYHA Class | 6 months
  NYHA Class Assessment
Change in quality of life score | 6 months
  Assessment through Minnesota Living with Heart Failure Questionnaire
Change in left ventricular ejection fraction | 6 months
  Improved left ventricular ejection fraction
Reduction in QRS duration | 6 months
  QRS duration measured on 12 lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Walton, BSc, Principal Investigator — University Hospitals Birmingham
Locations (1):
- University Hospitals Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No